CLINICAL TRIAL: NCT06076356
Title: Effects of Foam Roller Versus KT Tape on Delayed Onset Muscle Soreness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01615 Maria Nawaz
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Delayed Onset Muscle Soreness
Keywords: DOMS; Foam Rolling; HIIT; Kinesio Taping; Resistance Training

STUDY DESIGN:
Intervention Model Description: Concurrent Parallel Randomized Clinical Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Foam Rolling Group
  Interventions: Other: Foam Rolling
- Group B (Active Comparator): Kinesio Taping Group
  Interventions: Other: Kinesio Taping

INTERVENTIONS:
Other: Foam Rolling — Foam Roller for 90 seconds over anterior (quadriceps) and posterior (hamstrings) aspect of thigh.
  Arms: Group A
Other: Kinesio Taping — Kinesio taping over anterior (quadriceps) and posterior (hamstrings) aspect of thigh.
  Arms: Group B

SUMMARY:
Objective of this study is to compare the effects of foam roller with KT tape on DOMS. The university going students will be divided in two groups, with one group receiving Kinesio Tape as intervention and other Foam Rolling as intervention. Pain and range of motion will be assessed before and after the intervention and the effects of both interventions will be compared.

DETAILED DESCRIPTION:
Delayed Onset Muscle Soreness (DOMS) is a common phenomenon experienced after unaccustomed or intense physical activity, characterized by muscle discomfort, pain, and reduced range of motion. Various interventions have been conducted to alleviate DOMS symptoms, including the use of foam rollers and Kinesiology Tape (KT tape).

This randomized controlled clinical trial aims to compare the effects of foam roller and KT tape interventions on reducing DOMS and improving muscle recovery. The participants would go for a single session of High Intensity Interval Training (HIIT) to induce DOMS. Group-A participants would receive KT taping afterwards, while Group-B participants would receive foam rolling as intervention. Their effect would be measured using Visual Analog Scale (VAS), Tenderness Grading Scale, Knee Range of Motion (ROM) and Vertical Jump Height. This study delves into the applications and potential benefits of KT tape and foam roller in managing DOMS, shedding light on their effectiveness and how they can contribute to enhancing post-exercise recuperation and overall well-being.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with normal BMI (18.5 to 25 Kg/m2)

Exclusion Criteria:

* Individuals with history of metabolic or musculoskeletal disease.
* Individuals with any recent acute injury.
* Athletes exercising regularly and regular gymnasium going individuals.

Ages: 18 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The participant eligibility is based on self-representation of gender identity.
Enrollment: 24 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Pain (VAS Score) | Baseline, after 24 hours, after 48 hours, and after 72 hours
  Pain will be measured using Visual Analog Scale (VAS) ranging from zero (0=no pain) to ten (10=worst pain).
Tenderness | Baseline, after 24 hours, after 48 hours, and after 72 hours
  Tenderness will be measured using Tenderness Grading Scale ranging from zero (0=no tenderness) to four (4=severe tenderness).

SECONDARY OUTCOMES:
Knee Range of Motion (Flexion) | Baseline, after 24 hours, after 48 hours, and after 72 hours
  Range of motion will be measured using Universal Goniometer
Vertical Jump Height | Baseline, after 24 hours, after 48 hours, and after 72 hours
  Vertical Jump Height will be measured using Vertec.

CONTACTS AND LOCATIONS:
Overall Officials: Noman Sadiq, MS-SPT, Principal Investigator — Riphah International University, Islamabad.
Locations (1):
- Riphah International University (RIU), Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No